CLINICAL TRIAL: NCT05118074
Title: Nova Max Creatinine and eGFR Meter System - Evaluation
Brief Title: Nova Max Creatinine and eGFR Meter System
Status: Completed | Type: Observational
Sponsor: Nova Biomedical (Industry)
Collaborators: South Florida Research Organization (Unknown); Charisma Medical and Research Center (Unknown); Excellence Medical Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: NB21-eGFR-NA-FDA
Record Dates: First submitted 2021-07-28; First posted 2021-11-11 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Diseases; Acute Kidney Injury
Keywords: eGFR; Creatinine; POCT
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Creatinine, eGFR — Compare diagnostic tests to reference methods

SUMMARY:
To assess the performance of the Nova Max Creatinine and eGFR assay in the hands of CLIA-Waived Point-of-Care users in at least three (3) distinct Point-of-Care clinical settings on venous, and capillary blood and compare the performance characteristics to a traceable laboratory reference method (the Siemens EXL creatinine determination).

To assess the Ease of Use of the Nova Max Creatinine and eGFR Meter System in the hands of the intended CLIA-Waived Point-of-Care users.

DETAILED DESCRIPTION:
This study is designed to evaluate the performance of the NM Meter when used by CLIAW operators in terms of both accuracy to an established reference method and precision. CLIAW operators will receive no training or prompting on how to use the NM Creatinine and eGFR Meter, operating only using the instructions found in printed labeling materials (IFU, QRG, packaging).

In determining the accuracy of the device, subjects will be tested using the NM Creatinine and eGFR Meter alongside a central laboratory reference method and the results will be compared to one another. This portion of the study is referred to as Method Comparison.

In determining the precision of the device, multiple creatinine determinations will be made with the NM Creatinine and eGFR meter using both stabilized control materials (testing over the course of 20 days) and venous whole blood specimens (tested over the course of a single day). The difference between the multiple test results will determine the device's level of precision. This portion of the study is referred to as Precision.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females (≥ 18 years of age)
2. CKD Stage 1 (healthy)
3. CKD Stages 2-4
4. Subjects willing and able to consent to participating in the study.
5. Subjects whose pre-screen creatinine and eGFR value, if performed, is deemed valuable to the study.

Exclusion Criteria:

1. Subjects unable to consent to participating in the study.
2. Subjects possessing a cognitive disorder or other condition, which, in the opinion of the investigator, would put the person at risk or seriously compromise the integrity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified via medical records for history of CKD or compromised kidney function and contacted to participate in this study. Study site personnel will provide details regarding the study (requirements, test procedure, subject rights) to obtain informed consent from the subject.
  Potential subjects will be screened using the protocol inclusion and/or exclusion criteria. Adult subjects (≥ 18 years of age) with creatinine levels spanning the entire AMR of the NM Creatinine and eGFR Meter will be recruited for the study.
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Analytical verification of Nova Max creatinine and eGFR meter system - Creatinine comparison | 20 days
  Nova Max creatinine and eGFR meter system, a point of care testing instrument is as effective as a reference laboratory method for Creatinine blood results in mg/dL
Analytical verification of Nova Max creatinine and eGFR meter system - eGFR comparison | 20 days
  Nova Max creatinine and eGFR meter system, a point of care testing instrument is as effective as a reference laboratory method for eGFR blood results in mL/min/1.73 m^2

CONTACTS AND LOCATIONS:
Overall Officials: Giralt Yanez, Principal Investigator — South Florida Research Organization; Eduardo Alvarez, Principal Investigator — Charisma Medical and Research Center; Jeremy Bleicher, Principal Investigator — Excellence Medical Research
Locations (3):
- United States (3):
  - South Florida Research Organization, Medley, Florida
  - Excellence Medical Research, Miami Gardens, Florida
  - Charisma Medical and Research Center, Miami Lakes, Florida

IPD SHARING:
Plan to Share IPD: No